CLINICAL TRIAL: NCT01108523
Title: Open Label Evaluation of the Effects of HP828-101 in the Management of Moisture Associated Skin Damage in Adults
Brief Title: Evaluation of Effects of HP828-101 for Moisture Associated Skin Damage
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Business decision
Sponsor: Healthpoint (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 828-101-09-017
Record Dates: First submitted 2010-04-20; First posted 2010-04-22 (Estimated); Results first posted 2013-12-06 (Estimated); Last update posted 2013-12-06 (Estimated); Status verified 2013-10

CONDITIONS: Skin Abnormalities
Keywords: Moisture Associated Skin Damage
MeSH Terms: conditions — Skin Abnormalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HP828-101 (Experimental): HP828-101 Experimental Formulation
  Interventions: Device: HP828-101

INTERVENTIONS:
Device: HP828-101

SUMMARY:
This study evaluates HP828 in the management of moisture associated skin damage after 15 days of use.

ELIGIBILITY:
Inclusion Criteria:

* - The informed consent document must be read, signed, and dated by the subject or the subject's legally authorized representative before conducting any study procedures or exams. In addition, the informed consent document must be signed and dated by the individual who consents the subject before conducting Visit 1. A photocopy of the signed informed consent document must be provided to the subject or subject representative, and the original signed document placed in the subject's chart. If the subject is unable to read or sign the informed consent, or unable to comprehend the information provided in the consent process, a legal guardian, decision making proxy, or next of kin must provide written consent, and if possible, subject must verbally assent to receiving an experimental treatment for their wound.
* Are 18 years of age or older, of either sex and of any race or skin type provided that their skin color, in the opinion of the Investigator, will not interfere with the study assessments.
* Are expected to remain in the Nursing Home or long-term acute-care (LTAC) for the duration of the study (15 days).
* Have moisture associated skin damage including denuded skin or ulceration, where:

  * the damage has been present for at least 2 days but less than 6 weeks
  * the area of denudation (target wound) measures greater than or equal to 2 and less than or equal to 64 cm2 in total area
  * the area of total damage may be greater than 64 cm2
* Are able to verbally respond to the Pre- and Post- Treatment Survey.
* Women of child-bearing potential may participate in the study if they have a negative urine pregnancy test and use adequate birth control, as determined by the Investigator.
* Are capable of maintaining adequate nutritional intake during the study

Exclusion Criteria:

* Have more than 64 cm2 of denuded area.
* Have a full-thickness target wound, or a full-thickness wound within 4 cm of any target wound area.
* Have clinical evidence of bacterial or fungal infection of the target wound area.
* Have, within the area of moisture damaged skin, any tunneling, sinus tracks, shear injury, arterial occlusive disease, or bony prominence or joint with the exception that target wounds may be over dorsal spinous processes, coccyx, ischial tuberosities, or sacroiliac joints.
* Are moribund, or have a severe burn, debilitating immunodeficiency disorder, significant hematologic disorder, metastatic malignancy, uncontrolled diabetes mellitus, or any medical conditions that, in the opinion of the Investigator, places the subject at risk for the study or incapable of healing.
* Are known to have acrodermatitis enteropathica (zinc deficiency).
* Are being treated currently with systemic steroids, immunosuppressive agents, radiation, or chemotherapy.
* Have been treated with enzymatic debridement to the target wound area within 2 days prior to enrollment.
* Have a known sensitivity to ingredients of HP828-101.
* Are using or have used another investigational agent (not including devices such as hearing aids, pace makers, etc.) within 30 days prior to Visit 1.
* The Medical Monitor may declare any subject ineligible for a valid medical reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2010-04; Primary Completion 2010-07 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Herbert B Slade, MD, Study Chair — Healthpoint; Neeta Nayak, MD, Principal Investigator — Golden Acres
Locations (1):
- Golden Acres, Dallas, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Male or female subjects, age ≥ 18 years old, who were receiving care in a Nursing Home or Long Term Acute Care Facility (LTAC) and who had qualifying moisture damaged skin, with denudation in the range of 2 to 64 cm x cm
Period: Overall Study
Arm/Group | HP828-101
Started | 7
Completed | 3
Not Completed | 4
Not completed — Protocol Violation | 4

BASELINE CHARACTERISTICS:
Arm/Group | HP828-101
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 6
Age Continuous [Mean (Standard Deviation); unit: years] | 74.9 (15.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Rating Scores of Skin Erythema, Skin Pallor, Skin Maceration, Skin Denudation at Day 15.
Time Frame: 15 Days
Arm/Group | HP828-101
Number analyzed (Participants) | 0

2. Secondary Outcome: Rating Scores of Skin Erythema, Skin Pallor, Skin Maceration, Skin Denudation at Day 4, 8, and 12. Proportion of Subjects With no Denuded Skin Area at Day 4, 8, 12, and 15. Pre- and Post-Treatment Surveys
Time Frame: 4, 8, 12, and 15 days
Arm/Group | HP828-101
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | HP828-101
Serious Adverse Events (participants affected / at risk) | 1/7
Other Adverse Events (participants affected / at risk) | 0/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HP828-101 (N=7)
Metastatic brain cancer (Nervous system disorders) | 1 (1) — Subject enrolled in study despite a prior diagnosis & treatment for metastatic malignancy; was placed on Hospice care after exit from study with diagnosis of metastatic cancer of brain. Investigator determined it was not related to test article.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less